CLINICAL TRIAL: NCT05662982
Title: Evaluation of the Northwestern University Subischial Socket for Persons With Transfemoral Amputation and Lower Mobility Levels
Brief Title: Sub-Ischial Socket for Transfemoral Amputation and Lower Mobility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Stefania Fatone, Professor, School of Medicine, University of Washington
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00015284; CDMRP-E03034.1a (Other Grant/Funding Number: Congressionally Directed Medical Research Programs); CDMRP-E03034.1b (Other Grant/Funding Number: Congressionally Directed Medical Research Programs)
Record Dates: First submitted 2022-12-12; First posted 2022-12-23 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Transfemoral Amputation
Keywords: prosthesis; prosthetic socket

STUDY DESIGN:
Intervention Model Description: Two independent groups will be assessed longitudinally over 40 weeks: one group will be assessed using only the standard of care ischial containment socket and the other group will receive the subischial socket.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention Group (Experimental): Participants will be assessed for 12 weeks in their usual ischial containment socket before receiving a subischial socket to be worn and assessed for 24 weeks.
  Interventions: Device: Northwestern University Flexible Subischial Suction Socket (NU-FlexSIS)
- Reference Group (No Intervention): Participants will be assessed for 40 weeks in their usual ischial containment socket. No intervention will be provided.

INTERVENTIONS:
Device: Northwestern University Flexible Subischial Suction Socket (NU-FlexSIS) — A custom-made prosthetic socket for transfemoral amputation that consists of proximal trimlines that do not interact with the pelvis.
  Arms: Intervention Group

SUMMARY:
The objective of this trial is to assess use and benefits of the subischial socket for persons with transfemoral amputation and lower mobility levels. Specifically, the investigators will evaluate whether the subischial socket improves comfort, socket wear time, mobility, participation, quality of life and satisfaction with device than the standard-of-care ischial containment socket.

DETAILED DESCRIPTION:
Prosthetic sockets that are currently used by persons with above-the-knee amputation (AKA) fit intimately with the thigh and pelvis, limiting hip motion and causing discomfort. Socket comfort while standing and sitting is of great importance to persons with lower limb amputation. Yet discomfort while sitting has been reported in 44% of persons with AKA. In those with AKA who are more sedentary, clinical observation indicates that socket discomfort in sitting results in less prosthesis wear time and less mobility with the prosthesis. Based on these observations, the investigators propose that improving socket comfort in persons with AKA who have lower mobility will increase the time spent wearing the socket, which will in turn increase mobility, and in turn again improve satisfaction with the prosthesis and overall quality-of-life. A new prosthetic socket design, the sub-ischial socket, which eliminates contact with the pelvis, has been developed with the intent of improving comfort and hip motion in people with AKA. In particular, sitting comfort has been highlighted as an advantage of this new socket design by early users. Therefore, the objective of this project is to assess use and benefits of the sub-ischial socket for persons with AKA and lower mobility levels. The investigators will evaluate whether the sub-ischial socket is more comfortable, improves prosthesis wear time, mobility, participation in society, satisfaction with device, skin-related quality-of-life, and health-related quality of life compared to the current standard-of-care socket design in persons with AKA and lower mobility levels. If a participant is eligible and enrolled into this study, participation would last about 10 months and would involve up to 8 in-person visits (for individuals receiving a new sub-ischial socket). Individuals receiving a new sub-ischial socket will also be asked to wear a step counter and temperature sensor and complete 11 remote survey assessments spread over the 10-month period of the study. Data will also be collected from a reference group of participants with transfemoral amputation and lower mobility levels who will not receive a sub-ischial socket. These participants will be assessed while wearing their clinically-provided, standard-of-care ischial containment socket. These participants will complete 8 remote survey assessments over a 10-month period.

ELIGIBILITY:
Inclusion Criteria:

1. Speak and read English;
2. Provision of signed and dated informed consent form;
3. Stated willingness to comply with all study procedures and availability for the duration of the study;
4. All sexes and genders age 18 years and older;
5. Have a unilateral transfemoral or knee disarticulation amputation and have used a prosthesis for 1 year or more;
6. Be classified by their prosthetist as being a Medicare Functional Classification Level of K2 (limited community ambulator);
7. Have never worn a sub-ischial socket;
8. Current IC socket and prosthesis must be well fitting and maintained; current socket must have pelvic weightbearing and/or containment;
9. Participant has no plans to change the knee or foot in the next 10 months;
10. Willingness to adhere to the monitoring and new socket regimen;
11. Have sufficient upper limb function to don liner and change sensors;
12. Access to necessary resources for participating in the study (i.e., computer, smartphone, internet access, telephone):
13. Be a Veteran (VA site only).

Exclusion Criteria (intervention group only):

1. Have a femoral length <5 inches;
2. Have a known silicone allergy;
3. Are unable to don or tolerate wearing a compressive liner;
4. Loss of metatarsal heads on contralateral limb;
5. Active malignancy;
6. Pregnancy;
7. Polytrauma that affects functional ability beyond that of a unilateral transfemoral amputation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Socket Comfort Score (SCS) | Change from week 12 to week 24 compared between Intervention and Reference Groups.
  Single item self-report measure to rate average socket comfort on an 11-point scale where 0 represents the most uncomfortable socket fit participant can imagine and 10 represents the most comfortable socket fit participant can imagine. Participants will rate their socket comfort in general, and while sitting, standing, and walking.

SECONDARY OUTCOMES:
Temperature sensor | Intervention group only: Baseline period weeks 0-12; Intervention period weeks 0-24.
  Temperature sensor measures and records temperature and time at variable intervals. The temperature sensor will be retrofit to the liner worn with the usual socket and installed in the liner worn with the sub-ischial socket so that wear time can be monitored for the entire study duration.
Step counter | Intervention group only: Baseline period weeks 0-4; Intervention period weeks 0-4 and 20-24.
  A step counter activity monitor is an ankle-worn, microprocessor-controlled, two-dimensional accelerometer that measures step counts and step rates per unit time.
Prosthesis Limb Users Survey-Mobility (PLUS-M) | All participants: Baseline period weeks 0, 4, 8, 12; Intervention group: Intervention period weeks 4, 8, 12, 16, 20, 24; Reference group: Monitoring period weeks 4, 12, 20, 24.
  12-item self-report instrument for measuring mobility of adults with lower limb amputation (i.e., the ability to move intentionally and independently from one place to another). Items are rated on a scale from 1-5, with 1 indicating participants are unable to do the task and 5 indicating that participants can do it without any difficulty. Total raw scores range from 12-60. Raw scores are converted to a T-score using a lookup table, and final scores range from 20.3 to 67.7 on the T-score metric. The higher the total score the better the mobility.
Activities-specific Balance Confidence (ABC) Scale | All participants: Baseline period weeks 0, 4, 8, 12; Intervention group: Intervention period weeks 4, 8, 12, 16, 20, 24; Reference group: Monitoring period weeks 4, 12, 20, 24.
  16-item self-report measure where individuals rate their balance confidence in performing various activities without losing balance or experiencing a sensation of unsteadiness. Items are rated on a scale from 0-4, with 0 representing no balance confidence and 4 representing complete balance confidence. Total scores are created by averaging across the 16 items, with total scores ranging from 0 to 4. The higher the total score, the better the balance confidence.
Prosthesis Evaluation Questionnaire (PEQ) Residual Limb Health | All participants: Baseline period weeks 0, 4, 8, 12; Intervention group: Intervention period weeks 0, 4, 8, 12, 16, 20, 24; Reference group: Monitoring period weeks 4, 12, 20, 24.
  6-item self-report measure where individuals rate severity of residual limb issues such as rashes, sores, or sweating. Items are rated on a scale from 0-10, with 0 indicating that a residual limb problem/issue is very bothersome and 10 indicating that it is not at all bothersome. Total score is created by averaging across the 6 items, with possible scores ranging from 0-10. The higher the total score, the better the residual limb health.
Roland-Morris Disability Questionnaire (RMDQ) | All participants: Baseline period weeks 0, 4, 8, 12; Intervention group: Intervention period weeks 0, 4, 8, 12, 16, 20, 24; Reference group: Monitoring period weeks 4, 12, 20, 24.
  24-item self-report questionnaire used to determine the level of disability due to low-back pain. Items are rated as yes or no, with yes indicating that the responder endorses the statement as describing them today. Total score possible is 0-24, with scores indicative of the number of statements endorsed. The higher the total score, the more disabling the low-back pain.
Patient-Reported Outcomes Measurement Information System (PROMIS) Ability to Participate in Social Roles | All participants: Baseline period weeks 0, 12; Intervention/Monitoring period weeks 4, 12, 24.
  4-item self-report measure to assess satisfaction with one's usual social roles in life's situations and activities. These roles may exist in marital relationships, parental responsibilities, work responsibilities and social activities. Items are rated on a scale of 1-5 with 1 indicating participants always experienced the issue and 5 being never. Total raw score possible is 4-20. The raw score is converted to a t-score that ranges from 27.5 to 64.2 on the T-score metric. A higher score indicates better ability to participate in social roles.
Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health-10 | All participants: Baseline period weeks 0, 12; Intervention/Monitoring period weeks 4, 12, 24.
  10-item self-report measure used to assess general domains of health and functioning including overall physical health, mental health, social health, pain, fatigue, and overall perceived quality of life. Nine items are rated on a scale of 1-5 with a variety of response options (e.g., poor to excellent or always to never). The lower the score the worse health across all 9 items. One item is rated on a scale of 0-10 with 0 being no pain and 10 being worst imaginable pain. Four of the 10 items are combined to create a global mental health raw score that ranges from 4 to 20. Similarity, four items are combined to create a global physical health raw score that also ranges from 4 to 20. Raw scores are converted to T-scores and higher scores indicate better mental or physical health. The remaining two items are used individually in analyses and are not included in the overall physical or mental health scores.
Patient-Reported Outcomes Measurement Information System (PROMIS) Depression | All participants: Baseline period weeks 0, 12; Intervention/Monitoring period weeks 4, 12, 24.
  4-item self-report measure used to assess depression. Items are rated on a scale of 1-5 with 1 indicating participants have never experienced the issue and 5 being always. Total raw scores range from 4-20 and are converted to T-scores using a lookup table. Final T-scores range from 41.0 to 79.4. A lower score indicates less depressive symptoms.
Orthotic and Prosthetic Users' Survey Satisfaction with Device (OPUS-SwD) | All participants: Baseline period weeks 0, 12; Intervention/Monitoring period weeks 4, 12, 24.
  9-item self-report measure to assess satisfaction with device in persons who use prostheses. Items are rated 1-5 with 1 indicating strongly disagree and 5 indicating strongly agree. Total score possible is 9-45. The higher the score the better the satisfaction with device. The raw scores are converted to Rasch Measures.
Charlson Comorbidity Index (CCI) | All participants: Baseline period week 0; Intervention/Monitoring period weeks 4, 24.
  11-item self-report measure that assesses the presence of common health conditions. Items are rated as yes or no, with yes indicating participants have the health condition. Total score possible is 0-11. The higher the score, the more comorbid conditions the individual has.
Falls | All participants: Baseline period weeks 0, 4, 8, 12; Intervention group: Intervention period weeks 0, 4, 8, 12, 16, 20, 24; Reference group: Monitoring period weeks 4, 12, 20, 24.
  Falls will be self-reported by participants at each assessment time point. Participants will be asked if they have fallen in the past 4 weeks. If the participant indicates that they have fallen, they will ask how many times they have fallen in the past 4 weeks, whether the fall resulted in an injury, and if applicable, type of injury and whether they sought medical attention for the fall.

OTHER OUTCOMES:
Amputee Mobility Predictor with Prosthesis (AMP-Pro) | Intervention group only: Baseline period week 0; Intervention period weeks 0, 20.
  21-item in-person performance-based measure that assesses mobility potential of people with a lower limb prosthesis that evaluates transfers, sitting and standing balance, and gait skills. Items are variably scored, and item scores can range from 0-1 to 0-5. Total score possible is 0-47. The higher the score, the higher the mobility category.
International Society for Prosthetics and Orthotics (ISPO) Minimum Data Set for lower-limb prosthesis users involved Research Studies | Intervention group: Baseline period week 0; Intervention period week 0. Reference Group: Baseline period week 0.
  Descriptive information about the participant and prosthesis will include all the variables recommended by ISPO in their data set for lower-limb prosthesis users involved in research studies. These include participant characteristics (eg, age, weight, amputation level, reason for amputation, time since amputation, prosthetic experience, residual limb shape categorization, residual limb sensation qualitative assessment, lower extremity joint range of motion, manual muscle testing of lower limb strength, previous history of gait training with a therapist, and assistive device use). The list also includes prosthesis characteristics: structural design of prosthesis, socket type, suspension, prosthetic foot, ankle, shank and knee components, and type of residual limb socks.

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Fatone, PhD, Principal Investigator — University of Washington
Locations (3):
- United States (3):
  - Minneapolis VA Health Care System, Minneapolis, Minnesota
  - Hanger Institute for Clinical Research and Education, Houston, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Data generated by this research will be made available to the research community and to the public via University of Washington ResearchWorks digital repository of scholarly work. Prior to sharing, data will be de-identified and redacted to reduce the risk of participant identification. Final research data will include the factual material necessary to document and support research findings such as the outcome measure results and participant characteristics upon which any accepted publications are based, it may include both raw data and derived variables. Documentation will also be provided regarding the procedures used to collect and analyze the data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be shared no later than the acceptance for publication of the main findings from the final dataset.
Access Criteria: ResearchWorks creates persistent URLs that will not change over time. A DOI can also be created. The URL or DOI will be included with all publications arising from this trial.

REFERENCES:
- [Background] Fatone S, Caldwell R. Northwestern University Flexible Subischial Vacuum Socket for persons with transfemoral amputation-Part 1: Description of technique. Prosthet Orthot Int. 2017 Jun;41(3):237-245. doi: 10.1177/0309364616685229. Epub 2017 Jan 17. PMID 28094686
- [Background] Caldwell R, Fatone S. Technique modifications for a suction suspension version of the Northwestern University Flexible Sub-Ischial Vacuum socket: The Northwestern University Flexible Sub-Ischial Suction socket. Prosthet Orthot Int. 2019 Apr;43(2):233-239. doi: 10.1177/0309364618798869. Epub 2018 Sep 17. PMID 30223715
- [Background] Fatone S, Caldwell R, Angelico J, Stine R, Kim KY, Gard S, Oros M. Comparison of Ischial Containment and Subischial Sockets on Comfort, Function, Quality of Life, and Satisfaction With Device in Persons With Unilateral Transfemoral Amputation: A Randomized Crossover Trial. Arch Phys Med Rehabil. 2021 Nov;102(11):2063-2073.e2. doi: 10.1016/j.apmr.2021.05.016. Epub 2021 Jun 29. PMID 34214499
- [Background] Fatone S, Stine R, Caldwell R, Angelico J, Gard SA, Oros M, Major MJ. Comparison of Ischial Containment and Subischial Sockets Effect on Gait Biomechanics in People With Transfemoral Amputation: A Randomized Crossover Trial. Arch Phys Med Rehabil. 2022 Aug;103(8):1515-1523. doi: 10.1016/j.apmr.2022.02.013. Epub 2022 Mar 13. PMID 35296398

DOCUMENTS (4):
  • Informed Consent Form: UW-Hanger Intervention Group ICF 2023-07-27 (2023-07-27): https://cdn.clinicaltrials.gov/large-docs/82/NCT05662982/ICF_000.pdf
  • Informed Consent Form: MVAHCS Intervention Group ICF 2024-07-25 (2024-07-25): https://cdn.clinicaltrials.gov/large-docs/82/NCT05662982/ICF_003.pdf
  • Informed Consent Form: UW-Hanger Reference Group ICF 2023-08-31 (2023-08-31): https://cdn.clinicaltrials.gov/large-docs/82/NCT05662982/ICF_001.pdf
  • Informed Consent Form: UW Reference Group ICF 2024-03-01 (2024-03-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT05662982/ICF_002.pdf